CLINICAL TRIAL: NCT03037697
Title: Efficacy of Axial Stability on Improving Gait and Balance Performance in Children With Dyskinetic Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Umm Al-Qura University (Other)
Responsible Party: Principal Investigator, Shamekh Mohamed El-Shamy, Associate Professor, Umm Al-Qura University
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: Umm Al-Qura University
Record Dates: First submitted 2017-01-12; First posted 2017-01-31 (Estimated); Last update posted 2021-02-26 (Actual); Status verified 2021-02

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TheraTogs Arm (Experimental): TheraTogs Arm The participating children will wear TheraTogs orthotic undergarment and strapping as preparatory stage without application of any exercise program with gradually increasing the worn time till reaching the 8 hours per day, to allow the children to become acclimated to the system+ Traditional treatment 3 months
  Interventions: Other: TheraTogs Arm; Other: Traditional Treatment
- Traditional Treatment Arm (Active Comparator): Traditional Treatment Arm
  1-Trunk control exercises 2-Core stability training 3-Proximal dynamic stability for the shoulder and pelvic girdles components. 4- Back and abdominal strengthening exercises 5- Standing exercises : - Standing alone gradually increase time. - Stride standing alone. - Step standing alone (other limb supported on wooden step then soft step and finally on small ball). - Standing on balance board
  3 months
  Interventions: Other: Traditional Treatment

INTERVENTIONS:
Other: TheraTogs Arm — TheraTogs Arm Received Soft Orthotic undergarments
  Other Names: Experimental
  Arms: TheraTogs Arm
Other: Traditional Treatment — Traditional treatment to Dyskinetic CP
  1- Trunk control exercises 2- Core stability training 3- Proximal dynamic stability for the shoulder and pelvic girdles components. 4- Back and abdominal strengthening exercises 5- Standing exercises : - Standing alone gradually increase time. - Stride standing alone. - Step standing alone (other limb supported on wooden step then soft step and finally on small ball). - Standing on balance board

SUMMARY:
The aim of this study will be to evaluate the effect of TheraTogs orthotic undergarment and strapping system on increasing axial stability that will reflect on improving balance and walking performance in children with dyskinetic cerebral palsy.

DETAILED DESCRIPTION:
The aim of this study will be to evaluate the effect of TheraTogs orthotic undergarment and strapping system on increasing axial stability that will reflect on improving balance and walking performance in children with dyskinetic cerebral palsy. Forty children with dyskinetic CP will be assigned randomly into two groups (A & B). Control group (A) will receive conventional rehabilitation program for postural correction 2 hours/3 sessions weekly/3 successive months. Study group (B) will receive conventional rehabilitation program as in group (A) in addition to wearing Thera Togs soft orthotic undergarment. Patients evaluation will be carried out before and after the intervention programs to assess gait and balance performance using Noraxons myo pressure plate and Biodex balance system.

ELIGIBILITY:
Inclusion Criteria:

* The levels of gross motor function will be selected between levels I and II according to Gross Motor Function Classification System (GMFCS); have the ability to walk 10 m independently without an orthosis; should be cognitively competent and able to understand and follow instructions; height will be more than 100 cm to fit with the Biodex balance equipment.

Exclusion Criteria:

* If participants use an assistive mobility device; GMFCS levels III, IV, and V; fixed contractures of lower limb musculature; hip dislocation; significant spinal deformities.

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline gait parameters at 3 months | Baseline and 3 months post-intervention
  Gait parameters will be evaluated for every child at baseline and 3 months post-intervention using the Pro-Reflex motion analysis system (Qualisys; Qualisys Inc, Goeteborg, Sweden).

SECONDARY OUTCOMES:
Change from baseline postural stability at 3 months | Baseline and 3 months post-intervention
  Postural stability will be evaluated at baseline and 3 months post-intervention using the Biodex Balance System (BBS) (Balance System SD, Shirely, NY, USA).

CONTACTS AND LOCATIONS:
Overall Officials: Shamekh M El-Shamy, Ph.D, Principal Investigator — Associate Professor
Locations (1):
- Maternity and Children Hospital, Mecca, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No